CLINICAL TRIAL: NCT02984982
Title: A Randomized, Open-label, Blinded Intravascular Ultrasound Analysis, Parallel Group, Multicenter Study to Evaluate the Effect of Praluent® (Alirocumab) on Coronary Atheroma Volume in Japanese Patients Hospitalized for Acute Coronary Syndrome With Hypercholesterolemia Not Adequately Controlled With Statin
Brief Title: Evaluation of Effect of Alirocumab on Coronary Atheroma Volume in Japanese Patients Hospitalized for Acute Coronary Syndrome With Hypercholesterolemia
Acronym: ODYSSEY J-IVUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALIROL08069; U1111-1184-8764 (Other: UTN)
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Hypercholesterolemia; Acute Coronary Syndrome
MeSH Terms: conditions — Hypercholesterolemia; Acute Coronary Syndrome | interventions — alirocumab; Atorvastatin; Rosuvastatin Calcium; Fenofibrate; Bezafibrate; Ezetimibe; Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Statin therapy (atorvastatin or rosuvastatin) will be administered with or without non-statin lipid modifying therapies (LMTs). Non-statin LMTs will be adjusted by physicians to achieve the LDL-C target level <100 milligrams per deciliter (mg/dL).
  Interventions: Drug: Atorvastatin; Drug: Rosuvastatin; Drug: Fenofibrate; Drug: Bezafibrate; Drug: Ezetimibe; Drug: Antiplatelets; Drug: Anticoagulants
- Alirocumab (Experimental): Alirocumab will be given subcutaneously every 2 weeks on top of stable dose statin therapy (atorvastatin or rosuvastatin) with or without stable dose non-statin LMTs.
  Interventions: Drug: Alirocumab SAR236553; Drug: Atorvastatin; Drug: Rosuvastatin; Drug: Fenofibrate; Drug: Bezafibrate; Drug: Ezetimibe; Drug: Antiplatelets; Drug: Anticoagulants

INTERVENTIONS:
Drug: Alirocumab SAR236553 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Other Names: Praluent
  Arms: Alirocumab
Drug: Atorvastatin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Rosuvastatin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Fenofibrate — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Bezafibrate — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Ezetimibe — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Antiplatelets — Pharmaceutical form: tablet or capsule
  Route of administration: oral
Drug: Anticoagulants — Pharmaceutical form: tablet or capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

To compare the efficacy of alirocumab (Praluent®) with standard of care (SoC) on coronary atheroma progression (percent change in normalized total atheroma volume [TAV]) after 9 months of treatment in participants who had acute coronary syndrome (ACS) within 4 weeks prior to randomization, with hypercholesterolemia treated with statin.

Secondary Objectives:

* To compare the efficacy of alirocumab (Praluent®) with SoC on secondary endpoints including absolute change in percent atheroma volume and normalized TAV after 9 months of treatment.
* To evaluate the efficacy of alirocumab (Praluent®) on low-density lipoprotein cholesterol (LDL-C), apolipoprotein B, triglycerides, non-high-density lipoprotein cholesterol and lipoprotein (a) after 9 months treatment.
* To evaluate the safety of alirocumab (Praluent®) including the occurrence of cardiovascular events (coronary heart disease death, non-fatal myocardial infarction, fatal and non-fatal ischemic stroke, unstable angina requiring hospitalization) throughout the study.

DETAILED DESCRIPTION:
The duration of study per participant was 9 months.

ELIGIBILITY:
Inclusion criteria :

* Participants hospitalized for ACS (Acute ST-segment elevation myocardial infarction [STEMI], Acute non-ST-segment elevation myocardial infarction [NSTEMI], and unstable angina.
* LDL-C >=100 mg/dL at ACS diagnosis.
* Participants who has stenosis with at least >50% stenosis angiographically within 1 week after the ACS onset, and has analyzable coronary intravascular Ultrasound image.
* Participants aged >=20 years old at ACS diagnosis.
* Negative Hepatitis B surface antigen, negative Hepatitis B core antibody, and negative Hepatitis C antibody. Or, negative Hepatitis B surface antigen, positive Hepatitis B core antibody, negative Hepatitis B deoxyribonucleic acid, and negative Hepatitis C antibody.
* Written informed consent.

Exclusion criteria:

* Participants who had previously treated with at least one dose of any anti-proprotein convertase subtilisin/kexin type 9 monoclonal antibody.
* Uncontrolled hypertension (multiple reading with systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) between ACS diagnosis and randomization visit.
* Known history of hemorrhagic stroke.
* Currently under treatment for cancer.
* Participants on LDL apheresis.
* Any clinically significant abnormality identified that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study or constrain endpoints assessment such as major systemic diseases, participants with short life expectancy.
* Considered by the Investigator or any sub-Investigator as inappropriate for this study for any reason, including:

  * Unable to meet specific protocol requirements, such as scheduled visits;
  * Investigator or any sub-Investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol, etc;
  * Presence of any other conditions (eg, geographic, social, etc.) actual or anticipated, that the Investigator feels would restrict or limit the participant's participation for the duration of the study.
* Laboratory findings measured within 4 weeks after the ACS diagnosis (positive serum or urine pregnancy test in females of childbearing potential).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (39):
- Japan (39):
  - Investigational Site Number 392026, Bunkyō City
  - Investigational Site Number 392022, Chiyoda-ku
  - Investigational Site Number 392032, Fujisawa-shi
  - Investigational Site Number 392004, Fukui-shi
  - Investigational Site Number 392007, Fukuoka
  - Investigational Site Number 392048, Fukuoka
  - Investigational Site Number 392008, Gifu
  - Investigational Site Number 392039, Hiroshima
  - Investigational Site Number 392028, Isehara-shi
  - Investigational Site Number 392036, Itabashi-ku
  - Investigational Site Number 392037, Itabashi-ku
  - Investigational Site Number 392024, Izumisano
  - Investigational Site Number 392013, Izunokuni-shi
  - Investigational Site Number 392020, Kawaguchi-shi
  - Investigational Site Number 392009, Kitakyushu-shi
  - Investigational Site Number 392034, Kitakyushu-shi
  - Investigational Site Number 392044, Kochi
  - Investigational Site Number 392002, Kumamoto
  - Investigational Site Number 392011, Kumamoto
  - Investigational Site Number 392003, Kurashiki-shi
  - Investigational Site Number 392018, Matsuyama
  - Investigational Site Number 392021, Morioka
  - Investigational Site Number 392017, Nagakute-shi
  - Investigational Site Number 392047, Nagaoka-shi
  - Investigational Site Number 392033, Okayama
  - Investigational Site Number 392006, Osaka
  - Investigational Site Number 392010, Osaka
  - Investigational Site Number 392045, Osaka
  - Investigational Site Number 392046, Osaka
  - Investigational Site Number 392015, Sagamihara-shi
  - Investigational Site Number 392019, Sakaishi
  - Investigational Site Number 392035, Sapporo
  - Investigational Site Number 392001, Tenri-shi
  - Investigational Site Number 392016, Toyoake-shi
  - Investigational Site Number 392025, Tsukuba
  - Investigational Site Number 392040, Tsukuba
  - Investigational Site Number 392005, Wakayama
  - Investigational Site Number 392027, Yokohama
  - Investigational Site Number 392043, Yokohama

IPD SHARING:
Plan to Share IPD: No
Not available for request.

REFERENCES:
- [Derived] Ako J, Hibi K, Tsujita K, Hiro T, Morino Y, Kozuma K, Shinke T, Otake H, Uno K, Louie MJ, Takagi Y, Miyauchi K. Effect of Alirocumab on Coronary Atheroma Volume in Japanese Patients With Acute Coronary Syndrome - The ODYSSEY J-IVUS Trial. Circ J. 2019 Sep 25;83(10):2025-2033. doi: 10.1253/circj.CJ-19-0412. Epub 2019 Aug 20. PMID 31434809
- [Derived] Ako J, Hibi K, Kozuma K, Miyauchi K, Morino Y, Shinke T, Tsujita K, Uno K, Kawabata Y, Hiro T. Effect of alirocumab on coronary atheroma volume in Japanese patients with acute coronary syndromes and hypercholesterolemia not adequately controlled with statins: ODYSSEY J-IVUS rationale and design. J Cardiol. 2018 Jun;71(6):583-589. doi: 10.1016/j.jjcc.2017.11.013. Epub 2018 Mar 30. PMID 29606415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 active centers in Japan. Overall 214 participants were screened between 15 November 2016 and 02 November 2017, of whom 8 were screen failure and 206 were randomized to either alirocumab arm or standard of care (SoC) arm.
Pre-assignment Details: Randomization was stratified by 'on statin therapy' or 'not on statin therapy' at the time of acute coronary syndrome (ACS) onset.
Groups:
- Standard of Care: During the study period, participants randomized to the SoC arm, in a non-blinded manner, received orally, stable dose of statin therapy (atorvastatin greater than or equal to [>=] 10 milligram per day [mg/day] or rosuvastatin >=5 mg/day) with optional dose adjustment (within the range approved by health authority). In participants receiving statin monotherapy, non-statin, non-proprotein convertase subtilisin kexin type 9 (non-PCSK9) inhibitor lipid modifying therapies (LMTs) could be added by the investigators, if low-density lipoprotein cholesterol (LDL-C) target level less than (<) 100 milligrams per deciliter (mg/dL) could not be achieved.
- Alirocumab: Alirocumab (Praluent®) 75 mg subcutaneous (SC) injection every 2 weeks (Q2W) on top of stable dose statin therapy (atorvastatin >=10 mg/day or rosuvastatin >=5 mg/day). Statin (atorvastatin >=10 mg/day or rosuvastatin >=5 mg/day) and non-statin LMTs were continued at the same doses after ACS diagnosis unless modifications were necessary. Alirocumab (Praluent®) dose was increased to 150 mg Q2W at Week 14, if the Week 12 LDL-C was >=100 mg/dL.
Period: Overall Study
Arm/Group | Standard of Care | Alirocumab
Started | 102 | 104
Treated | 102 | 103
Completed | 94 | 94
Not Completed | 8 | 10
Not completed — Adverse Event | 2 | 5
Not completed — Poor Compliance to Protocol | 4 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants who were allocated to a randomized treatment and recorded in the registration center database, regardless of whether a study drug was used or not.
Groups:
- Standard of Care: During the study period, participants randomized to the SoC arm, in a non-blinded manner, received orally, stable dose of statin therapy (atorvastatin >=10 mg/day or rosuvastatin >=5 mg/day) with optional dose adjustment (within the range approved by health authority). In participants receiving statin monotherapy, non-statin, non-PCSK9 inhibitor LMTs could be added by the investigators, if LDL-C target level <100 mg/dL could not be achieved.
- Alirocumab: Alirocumab (Praluent®) 75 mg SC injection Q2W on top of stable dose statin therapy (atorvastatin >=10 mg/day or rosuvastatin >=5 mg/day). Statin (atorvastatin >=10 mg/day or rosuvastatin >=5 mg/day) and non-statin LMTs were continued at the same doses after ACS diagnosis unless modifications were necessary. Alirocumab (Praluent®) dose was increased to 150 mg Q2W at Week 14, if the Week 12 LDL-C was >=100 mg/dL.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Alirocumab | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.9) | 61.7 (10.9) | 60.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 83 | 83 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 102 | 104 | 206
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - high density lipoprotein [HDL] cholesterol - [Triglycerides/5]). Population: "Number analyzed" = Number of participants evaluable for the specified baseline measure.
  mg/dL
    number analyzed (Participants) | 98 | 103 | 201
    (all) | 95.2 (22.6) | 98.5 (22.9) | 96.9 (22.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Normalized Total Atheroma Volume (TAV) at Week 36
Description: Least-squares (LS) means and standard errors (SE) at Week 36 were obtained from analysis of covariance (ANCOVA) model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and the baseline normalized TAV as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: Modified intent-to-treat (mITT) population: all participants who were allocated to a randomized treatment, recorded in the registration center database, had at least one dose or part of dose of study drug and had 2 analyzable normalized TAV values, 1 assessed before randomization, and one assessed after 24 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | -3.14 (0.97) | -4.79 (0.95)
Statistical Analysis 1: Comparison: Standard of Care vs Alirocumab; Analysis was performed using ANCOVA model which included fixed categorical effects of treatment arm and randomization strata, as well as the continuous fixed covariate of baseline normalized TAV; Test type: Superiority; p = 0.2279, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -1.64, 95% CI 2-sided [-4.32 to 1.04], Standard Error of Mean 1.36 — Standard of Care vs Alirocumab

2. Secondary Outcome: Absolute Change From Baseline in Percent Atheroma Volume (PAV) at Week 36
Description: LS mean and SE at Week 36 were obtained from ANCOVA model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and the baseline PAV as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent atheroma volume
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent atheroma volume | -1.28 (0.39) | -1.42 (0.38)

3. Secondary Outcome: Absolute Change From Baseline in Normalized Total Atheroma Volume at Week 36
Description: LS mean and SE at Week 36 were obtained from ANCOVA model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and the baseline normalized TAV as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: cubic millimeter (mm^3)
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
cubic millimeter (mm^3) | -4.73 (1.02) | -5.77 (1.00)

4. Secondary Outcome: Absolute Change From Baseline in External Elastic Membrane (EEM) Volume at Week 36
Description: Adjusted mean and SE at Week 36 were obtained from robust regression model with treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]), as fixed categorical effects, and the baseline EEM volume value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mm^3 | -8.23 (1.85) | -10.01 (1.81)

5. Secondary Outcome: Percent Change From Baseline in External Elastic Membrane Volume at Week 36
Description: Adjusted mean and SE at Week 36 were obtained from robust regression model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and the baseline EEM volume value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Standard of Care: During the study period, participants randomized to the SoC arm, in a non-blinded manner, received orally, stable dose of statin therapy (atorvastatin >=10 milligram per day [mg/day] or rosuvastatin >=5 mg/day) with optional dose adjustment (within the range approved by health authority). In participants receiving statin monotherapy, non-statin, non-PCSK9 inhibitor lipid modifying therapies (LMTs) could be added by the investigators, if LDL-C target level <100 mg/dL could not be achieved.
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | -0.86 (0.93) | -3.18 (0.91)

6. Secondary Outcome: Absolute Change From Baseline in Lumen Volume at Week 36
Description: Adjusted mean and SE at Week 36 were obtained from robust regression model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and the baseline lumen volume value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mm^3 | -1.25 (1.38) | -0.93 (1.35)

7. Secondary Outcome: Percent Change From Baseline in Lumen Volume at Week 36
Description: Adjusted mean and SE at Week 36 were obtained from robust regression model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effect, and the baseline lumen volume value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: mITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | 1.20 (1.26) | -0.86 (1.23)

8. Secondary Outcome: Absolute Change From Baseline in Calculated Low-density Lipoprotein Cholesterol at Week 12 and Week 36
Description: Adjusted LS mean and SE at Week 12 and Week 36 were obtained from mixed-effect model including all available post-baseline data from Week 4 to Week 36. Model included treatment arm (SoC arm, alirocumab arm), randomization strata (statin at ACS onset [Yes / No]), time point, treatment-by-time point and randomization strata-by-time point interaction as fixed categorical effects, and baseline calculated LDL-C value and baseline calculated LDL-C value-by-time point interaction as continuous fixed covariates.
Time Frame: Baseline, Week 12, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline calculated LDL-C values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 85 | 93
mg/dL
  Week 12 | -9.6 (1.7) | -62.4 (1.6)
  Week 36 | -15.5 (1.8) | -63.2 (1.8)

9. Secondary Outcome: Percent Change From Baseline in Calculated Low-density Lipoprotein Cholesterol at Week 12 and Week 36
Description: as for outcome 8
Time Frame: Baseline, Week 12, Week 36
Population: mITT population with one baseline and at least one post-baseline calculated LDL-C values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 85 | 93
percent change
  Week 12 | -7.57 (1.91) | -64.53 (1.83)
  Week 36 | -13.40 (1.99) | -63.94 (1.91)

10. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B (Apo B) at Week 36
Description: Adjusted LS mean and SE at Week 36 were obtained from ANCOVA model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and baseline Apo B value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and one post-baseline Apo B values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
mg/dL | -16.8 (1.4) | -51.0 (1.3)

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 36
Description: as for outcome 10
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and one post-baseline Apo B values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
percent change | -16.61 (1.56) | -55.13 (1.53)

12. Secondary Outcome: Absolute Change From Baseline in Non-High-density Lipoprotein Cholesterol (Non-HDL-C) at Week 36
Description: Adjusted LS mean and SE at Week 36 were obtained from mixed-effect model including all available post-baseline data from Week 4 to Week 36. Model included treatment arm (SoC arm, alirocumab arm), randomization strata (statin at ACS onset [Yes / No]), time point, treatment-by-time point and randomization strata-by-time point interaction as fixed categorical effects, and baseline calculated non-HDL-C value and baseline calculated non-HDL-C value-by-time point interaction as continuous fixed covariates.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mg/dL | -20.3 (2.0) | -69.2 (2.0)

13. Secondary Outcome: Percent Change From Baseline in Non-High-density Lipoprotein Cholesterol at Week 36
Description: as for outcome 12
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | -14.06 (1.71) | -54.50 (1.67)

14. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol (TC) at Week 36
Description: LS mean and SE at Week 36 were obtained from mixed-effect model including all available post-baseline data from Week 4 to Week 36. Model included treatment arm (SoC arm, alirocumab arm), randomization strata (statin at ACS onset [Yes / No]), time point, treatment-by-time point and randomization strata-by-time point interaction as fixed categorical effects, and baseline calculated TC value and baseline calculated TC value-by-time point interaction as continuous fixed covariates.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline TC values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mg/dL | -15.2 (2.3) | -61.7 (2.2)

15. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 36
Description: Adjusted LS mean and SE at Week 36 were obtained from mixed-effect model including all available post-baseline data from Week 4 to Week 36. Model included treatment arm (SoC arm, alirocumab arm), randomization strata (statin at ACS onset [Yes / No]), time point, treatment-by-time point and randomization strata-by-time point interaction as fixed categorical effects, and baseline TC value and baseline TC value-by-time point interaction as continuous fixed covariates.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline TC values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | -7.59 (1.35) | -35.43 (1.32)

16. Secondary Outcome: Absolute Change From Baseline in Lipoprotein (a) (Lp[a]) at Week 36
Description: Adjusted mean and SE at Week 36 were obtained from robust regression model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effect, and baseline Lp(a) value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and post-baseline Lp(a) values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
mg/dL | -10.3 (0.5) | -15.5 (0.5)

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 36
Description: as for outcome 16
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and one post-baseline Lp(a) values.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
percent change | -17.23 (2.60) | -55.76 (2.54)

18. Secondary Outcome: Absolute Change From Baseline in High-density Lipoprotein Cholesterol at Week 36
Description: Adjusted LS mean and SE at Week 36 were obtained from mixed-effect model including all available post-baseline data from Week 4 to Week 36. Model included treatment arm (SoC arm, alirocumab arm), randomization strata (statin at ACS onset [Yes / No]), time point, treatment-by-time point and randomization strata-by-time point interaction as fixed categorical effects, and baseline HDL-C value and baseline HDL-C value-by-time point interaction as continuous fixed covariates.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline HDL-C values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mg/dL | 4.7 (0.9) | 8.1 (0.9)

19. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol at Week 36
Description: as for outcome 18
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline HDL-C values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | 12.19 (2.30) | 21.04 (2.25)

20. Secondary Outcome: Absolute Change From Baseline in Fasting Triglycerides (TGs) at Week 36
Description: Adjusted mean and SE were obtained from multiple imputation approach followed by robust regression model including fixed categorical effect of treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) and the continuous fixed covariate of baseline fasting TGs value.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline fasting TGs values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
mg/dL | -26.2 (4.7) | -35.3 (4.5)

21. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 36
Description: Adjusted mean and SE were obtained by multiple imputation approach followed by robust regression model included fixed categorical effect of treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) and the continuous fixed covariate of baseline fasting TGs value.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and at least one post-baseline fasting TGs values.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 89 | 93
percent change | -8.85 (3.62) | -18.37 (3.51)

22. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 36
Description: Adjusted LS mean and SE at Week 36 were obtained from ANCOVA model including treatment arm (SoC arm, alirocumab arm) and randomization strata (statin at ACS onset [Yes / No]) as fixed categorical effects, and baseline Apo A-1 value as continuous fixed covariate.
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and one post-baseline Apo A-1 values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
mg/dL | 3.8 (1.9) | 12.0 (1.9)

23. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 at Week 36
Description: as for outcome 22
Time Frame: Baseline, Week 36
Population: Participants of the mITT population with one baseline and one post-baseline Apo A-1 values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 88 | 92
percent change | 4.61 (1.62) | 11.75 (1.58)

24. Secondary Outcome: Number of Participants With Cardiovascular (CV) Adverse Events
Description: The suspected or confirmed CV events that occurred from randomization until end of the study visit were collected and reported. The various CV events included CV death, myocardial infarction, ischemic stroke, unstable angina requiring hospitalization , congestive heart failure requiring hospitalization, congestive heart failure requiring hospitalization, ischemia-driven coronary revascularization procedure.
Time Frame: Up to 36 weeks
Population: Safety population: all participants who actually received at least 1 dose or part of a dose of the study drug, and analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Alirocumab
Number analyzed (Participants) | 102 | 103
Participants
  Cardiovascular death | 0 | 0
  Myocardial infarction | 3 | 2
  Ischemic stroke | 0 | 2
  Unstable angina requiring hospitalization | 0 | 0
  Congestive heart failure requiring hospitalization | 0 | 0
  Ischemia led coronary revascularization procedure | 2 | 4

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to 21 days after last dose of study drug, or end of study, whichever comes first (up to 39 weeks) regardless of seriousness or relationship to investigational product
Description: Reported AEs and deaths are treatment-emergent adverse events that developed/worsened during the treatment-emergent period (time from first dose of investigational medicinal product (IMP) up to last dose of IMP +21 days, or end of study, whichever comes first). Analysis was performed on safety population.
Arm/Group | Standard of Care | Alirocumab
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/103
Serious Adverse Events (participants affected / at risk) | 17/102 | 19/103
Other Adverse Events (participants affected / at risk) | 15/102 | 33/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=102) | Alirocumab (N=103)
Anal abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=102) | Alirocumab (N=103)
Nasopharyngitis (Infections and infestations) | 15 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Injection site reaction (General disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT02984982/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT02984982/SAP_001.pdf